CLINICAL TRIAL: NCT00933361
Title: Individual Dose-escalated Bi-daily sc Ghrelin in Cancer Cachexia: a Phase I/II Study
Brief Title: Individual Dose-escalated Bi-daily Subcutaneously (sc) Ghrelin in Cancer Cachexia: a Phase I/II Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Bachem (Other)
Responsible Party: Principal Investigator, Florian Strasser, MD ABHPM, Associate Professor Clinic for Oncology and Hematology, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG 294/08
Record Dates: First submitted 2009-07-06; First posted 2009-07-07 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Advanced Cancer; Cachexia
Keywords: Adult
MeSH Terms: conditions — Cachexia | interventions — Ghrelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ghrelin (Experimental): Ghrelin, a 28 amino acid peptide discovered in 1999, is predominantly secreted by gastric endocrine cells and is an endogenous ligand for the growth hormone secretagogue (GHS) receptor. When administered peripherally it stimulates growth hormone secretion, food intake, triggers a positive energy balance, produces weight gain through a central mechanism involving hypothalamic neuropeptides and has anti-inflammatory effects
  Interventions: Drug: ghrelin

INTERVENTIONS:
Drug: ghrelin — As starting dose the investigators choose a dose level which was shown in our last study to be safe in human beings, i.e. 8μg/kg intravenously. With an assumed bioavailability of 25% of subcutaneously administered ghrelin the corresponding dose for dose level 1 is therefore 32 μg/kg. In the first 4 dose levels for each subsequent dose level the dose is increased by 50% compared to the previous one, from the 5th dose level onwards the increase is 25%: Dose level 1 = 32 μg/kg Dose level 2 = 48 μg/kg Dose level 3 = 72 μg/kg Dose level 4 = 108 μg/kg Dose level 5 = 135 μg/kg Dose level 6 = 169 μg/kg Dose level 7 = 211 μg/kg The investigators define the maximum tolerable dose as 20mg ghrelin (equivalent to 5ml) for reasons of the high drug volume to be administered subcutaneously.

SUMMARY:
Cachexia, a condition of severe malnutrition, negative nitrogen balance, muscle wasting, weight loss, and anorexia, is a frequent affecting more than 80% of patients in advanced cancer disease causing a high burden on patients and their families. Nutritional, pharmacological, and behavioural interventions for cancer-related ACS and associated symptoms have, despite the importance for cancer care, limited effect on only a minority of patients. New strategies are required.

Ghrelin, a 28 amino acid peptide discovered in 1999, is predominantly secreted by gastric endocrine cells and is an endogenous ligand for the growth hormone secretagogue (GHS) receptor. When administered peripherally it stimulates growth hormone secretion, food intake, triggers a positive energy balance, produces weight gain through a central mechanism involving hypothalamic neuropeptides and has anti-inflammatory effects. A recently completed trial on intravenous ghrelin in advanced cancer patients with ACS reports good tolerability and safety of single intravenous application of 2 and 8μg/kg Ghrelin.

Given the facts that ACS is a major burden in patients suffering advanced cancer disease and ghrelin is a major signal for stimulating food intake, promoting positive energy balance and weight gain and may have anti-inflammatory effect it remains to be determined whether the administration of ghrelin will have a positive clinical effect on cancer anorexia/ cachexia syndrome ACS. The next logical clinical development step is a proper dose-finding study of twice daily subcutaneous administration and proof-of-concept of main outcomes.

ELIGIBILITY:
Inclusion:

* Age: Patients must be older than 18 years of age
* Tumour situation: Patients with any type of advanced (defined as locally recurrent or metastatic), incurable solid tumour.
* Cachexia: defined as involuntary loss of weight of ≥2% in 2 months or ≥5% in 6 months, and ongoing in the last 4 weeks
* No simple starvation: Patients must be able to eat, defined as no severe structural barriers in the upper gastrointestinal tract and no bowel obstruction.
* No late cachexia: Patient must have an expected life expectancy > 3 months
* No anti-cachexia or appetite-stimulating medications: Patients are not allowed to have corticosteroids unless for maximum 2 days for chemotherapy, no progestin therapy within the last 2 weeks, no anabolic drugs within the last month. Prokinetic medication, NSAR (paracetamol and novamin sulphate are allowed, if given in a fixed dose for two weeks before visit 1, and expected to be given during the whole trial period.
* Laboratory test results within these ranges: Absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, serum creatinine ≤ 2.0 mg/dL (177 μmol/L), creatinine clearance ClCr ≥ 50ml/min, total bilirubin ≤1.5 mg/dL (25μmol/L), and AST (SGOT)/ ALT (SGPT) ≤2 x ULN or if hepatic metastases are present ≤ 5 x ULN.
* No other trial: Patient is not or was not participating in any other clinical trial within 28 before visit 2.
* Women of childbearing potential: A negative pregnancy test & effective contraception are mandatory in child-bearing age.
* Men agree not to father a child (i.e. use adequate birth control if sexually active) during participation in the trial.
* Cognition: Presence of a normal level of consciousness (mandatory is a normal abbreviated screening mini-mental test or a common mini-mental ≥ 27/30; in elderly patients age ≥ 65 years or patients with low education a mini mental status of ≥25/30 points will be considered adequate).
* Consent: The patient has voluntarily signed and dated an independent Ethics Committee (IEC) approved consent prior to any study-specific procedures.
* Gastrectomy: Patients with history of gastrectomy are eligible.

Exclusion:

* Questionnaires: Any psychiatric disorder, alcohol and illicit drug abuser language problem that would prevent the patient from filling in the questionnaires adequately.
* Patient with a history of psychiatric diagnosis of depression or clinical diagnosis of depression as determined by the treating physician or Hospital Anxiety Depression Scale total score of 13 or greater.
* History of alcohol abuse as determined by the CAGE questionnaire (≥2/4) or history of illicit drug abuse within last 12 months.
* Parenteral nutrition
* Diabetes mellitus with secondary organ dysfunction: coronary heart disease, previous stroke, renal insufficiency
* Patients with cerebral metastases or prophylactic whole brain irradiation for possible cerebral metastases.
* Known hypersensitivity to ghrelin.
* Known infection with HIV or a viral hepatitis
* Patients with known myeloid malignancy or tumours having bone marrow involvement
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the dose of ghrelin in tumour patients with ACS causing optimal stimulation of nutritional intake - minimal dose for maximal nutritional intake (MD-MANI) - or the maximally tolerable dose (MTD), which one occurs first | bi-weekly
To assess the effect of ghrelin on muscle strength. | weekly

SECONDARY OUTCOMES:
To assess the toxicity and tolerability, pharmacokinetics and symptoms of eating of ghrelin. | bi-weekly
To assess the effect of ghrelin on muscle mass, physical function, safety, toxicity and tolerability, pharmacokinetics, symptoms of eating, gastrointestinal motility, inflammation | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Florian Strasser, PD Dr. MD, Principal Investigator — Cantonal Spital St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen KSSG, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Strasser F, Lutz TA, Maeder MT, Thuerlimann B, Bueche D, Tschop M, Kaufmann K, Holst B, Brandle M, von Moos R, Demmer R, Cerny T. Safety, tolerability and pharmacokinetics of intravenous ghrelin for cancer-related anorexia/cachexia: a randomised, placebo-controlled, double-blind, double-crossover study. Br J Cancer. 2008 Jan 29;98(2):300-8. doi: 10.1038/sj.bjc.6604148. Epub 2008 Jan 8. PMID 18182992